CLINICAL TRIAL: NCT05798052
Title: Managing Medical Crisis - The Effects of Stress on Team Communication, Coordination and Performance
Brief Title: Effects of Stress on Team Coordination and Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020752-01H
Record Dates: First submitted 2023-03-08; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Stress Reaction; Stress, Psychological; Stress, Physiological
Keywords: teamwork; coordination
MeSH Terms: conditions — Fractures, Stress; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Teams will be assigned to manage simulated clinical scenarios in two order: low stress then high stress, high stress then low stress.
Who Masked: Outcomes Assessor
Masking Description: Assessors, who are blinded to the study hypotheses and manipulations, will score video-recordings of the teams, in terms of their performance and their coordination patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-High stress group (Other): Complete the first simulated clinical scenario in the low stress condition, then complete the second simulated scenario in the high stress condition.
  Interventions: Behavioral: Psychological stressors added to simulated clinical scenarios.
- High-Low stress groups (Other): Complete the first simulated clinical scenario in the high stress condition, then complete the second simulated scenario in the low stress condition.
  Interventions: Behavioral: Psychological stressors added to simulated clinical scenarios.

INTERVENTIONS:
Behavioral: Psychological stressors added to simulated clinical scenarios. — In both low and high stress scenario versions, the underlying mechanism of disease or injury will be identical, as will be the expected clinical management of the situation. Known stressors9,10 will be added to the scenarios, ensuring ecological validity (stressors that occur in real life). The stressors will include a) socio-evaluative stressors (presence of other with ability to negatively judge); b) increases in the severity of the situation (unstable patient); c) increases in the stakes (e.g. woman in early stages of pregnancy), d) noise, as well as e) unexpected brief complications (e.g. brief equipment challenge).

SUMMARY:
Healthcare teams often encounter challenging circumstances where they must deliver high-quality care. For a team to function effectively, its members must not only be individually competent, but they also need to collaborate and cooperate using their respective expertise. Such teams often work under high stress situations, where they need to make high stakes decisions under conditions of uncertainty, time-sensitivity and variable levels of control. Research shows that such emergency situations provoke stress responses in individuals, which can impair attention, memory, reasoning, and decision-making. However, it remains unclear how individual-level stress responses influence team communication, coordination, and performance. The aims of this study are to a) compare team coordination, communication, and performance in low stress versus high stress simulated emergency situations; and b) characterize the relationship between teams' stress profiles and the teams' performance and coordination. The study will be a within-subject experimental design, with teams serving as their own controls. Teams of emergency medicine residents and nurses will participate in two simulation scenarios: one in a low stress condition, and the other in a high stress condition (counterbalanced across the teams).

DETAILED DESCRIPTION:
Healthcare teams often encounter challenging circumstances where they must deliver high-quality care. For a team to function effectively, its members must not only be individually competent, but they also need to collaborate and cooperate using their respective expertise. Effective teamwork has been demonstrated to have a positive effect on patient outcomes and adherence to treatment guidelines. As a result, team training interventions have become increasingly prevalent in healthcare. These interventions predominantly focus on generic team competencies that can be transported across different situations and team compositions. A recent meta-analysis found that team training resulted in large effect sizes for the learning and transfer of cognitive and skills-based outcomes, but weaker effects on teamwork performance and medical errors. As such, there are calls to better understand the factors that affect teamwork. Teams often work under high stress situations, where they need to make high stakes decisions under conditions of uncertainty, time-sensitivity and variable levels of control. Research shows that such emergency situations provoke stress responses in individuals, which can impair attention, memory, reasoning, and decision-making. However, it remains unclear how individual-level stress responses influence team communication, coordination, and performance. The aims of this study are to a) compare team coordination, communication, and performance in low stress versus high stress simulated emergency situations; and b) characterize the relationship between teams' stress profiles and the teams' performance and coordination.

Methods: The study will be a randomized control trial, with teams serving as their own controls. Teams of emergency medicine residents and nurses will participate in two simulation scenarios: one in a low stress condition, and the other in a high stress condition (counterbalanced across the teams). Based on previous similar studies on the impact of stress on individual performance, where large effects sizes are seen (.7 -.75)8, the study will recruit a minimum of 17 teams (two-tailed test, alpha set at .05 and power set at .80). In both low and high stress scenario versions, the underlying mechanism of disease or injury will be identical, as will be the expected clinical management of the situation. Known stressors will be added to the scenarios, ensuring ecological validity (stressors that occur in real life). The stressors will include a) socio-evaluative stressors (presence of other with ability to negatively judge); b) increases in the severity of the situation (unstable patient); c) increases in the stakes (e.g. woman in early stages of pregnancy), d) noise, as well as e) unexpected brief complications (e.g. brief equipment challenge).

The participants' subjective (State-Trait Anxiety Inventory- STAI11, cognitive appraisal) and physiological stress (heart rate variability) responses will be measured. Stress responses will be compared at baseline, immediately before, and immediately after each scenario, as well as during for the physiological measures. The team performance will be assessed using the Team Emergency Assessment Measure (TEAM).

ELIGIBILITY:
Inclusion Criteria:

* Teams of postgraduate residents enrolled at the University of Ottawa, and The Ottawa Hospital emergency medicine nurses scheduled to attend simulation education sessions organized within their department.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Team performance | Over 3 months at the end of the data collection phase.
  Team performance will be assessed using the Team Emergency Assessment Measure (TEAM), which was developed to assess the quality of medical emergency team performance. It consists of 12 items. The first 11 items assess leadership, team coordination, team communication, and situation awareness on 5-point Likert scale. The 12th item is an overall measure of a team's performance and scored on a 10-point Likert-scale. Higher scores indicate better performance. The teams performance during the scenarios will be video-recorded and then scored by blinded raters

SECONDARY OUTCOMES:
Ratio of information management to task management | Over 3 months at the end of the data collection phase.
  Using a structured observation system of team coordination during non-routine events (Co-ACT, Framework for Observing Coordination Behaviour in Acute Care Teams), the investigators will characterize how and when the teams engage in coordination and communication activities that have been linked with high performing teams, but that have yet to be integrated into common healthcare team training approaches. The ratio of information management versus task management will be calculate as the amount of time in which the team members communicate and coordinate actions related to information management versus the amount of time communicating and coordinating actions related to task management. The teams performance during the scenarios will be video-recorded and then scored by blinded raters
Frequency of chances between implicit and explicit coordination | Over 3 months at the end of the data collection phase.
  Using a structured observation system of team coordination during non-routine events (Co-ACT, Framework for Observing Coordination Behaviour in Acute Care Teams), the investigators will characterize how and when the teams engage in coordination and communication activities that have been linked with high performing teams, but that have yet to be integrated into common healthcare team training approaches. The frequency of changes between implicit coordination and explicit coordination will be calculated as the number of times, in a given scenario, the team switches from implicit coordination to explicit coordination, and vice-versa. The teams performance during the scenarios will be video-recorded and then scored by blinded raters,
Team heedfulness score | Over 3 months at the end of the data collection phase.
  Using a structured observation system of team coordination during non-routine events (Co-ACT, Framework for Observing Coordination Behaviour in Acute Care Teams), the investigators will characterize how and when the teams engage in coordination and communication activities that have been linked with high performing teams, but that have yet to be integrated into common healthcare team training approaches. The degree of heedfulness in the teams will be calculated as the total time that team members engage in heedful behaviours (Noticing and communicating, Anticipating, Maintaining standards, Backup Behaviour, Closed-Loop Communication). The teams performance during the scenarios will be video-recorded and then scored by blinded raters

OTHER OUTCOMES:
Subjective Stress responses | Through study completion, and average of 1 year
  As a manipulation check, the investigators will compare the team subjective stress scores between the low stress and high stress scenarios. Subjective stress will be assessed with the Y Form of the State-Trait Anxiety Inventory (STAI), a 20-item tool designed to measure an individual's momentary level of anxiety by self-report. The STAI has been shown to be sensitive to manipulations of acute stress in simulated settings. Each inventory is scored between 20 and 80, and has population anxiety reference ranges available. Higher scores indicate greater levels of anxiety. In this study, participants will complete the STAI at baseline, immediately before, and immediately after each scenario.
Cognitive appraisal | Through study completion, an average of 1 year
  As a manipulation check, cognitive appraisal will be assessed immediately before and after each scenario. Primary appraisal will be examined by asking the participants to answer the questions 'How demanding do you expect the upcoming task to be?' before the scenario and 'How demanding was the task you just completed?' after the scenario. Secondary appraisal will be measured by asking the participants to answer the question: 'How able are [were] you to cope with this task?' Participants will indicate their answers on an anchored 10-point Likert scale. The index of cognitive appraisal is calculated as the ratio of the primary appraisal (demands) to the secondary appraisal (resources). If the resources are assessed as being equal to or greater than the task demands, the situation is appraised as a 'challenge' (ratio ≤ 1). If the task demands are appraised as being greater than the resources, the situation is appraised as a 'threat' (ratio > 1). I
Heart rate variability - rMSSD | During the simulation sessions, throughout the study: 5 minutes at start of each session (Baseline), 5 minutes prior to start of each scenario, for the duration of each scenario (divided into sequential 5 min periods), 5 minutes following each scenario
  As manipulation check, the investigators will compare the team physiological stress scores between the low stress & high stress scenarios by heart rate variability (HRV) monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants HRV will be recorded for 5 minutes at the start of the session (Baseline), 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of each scenario (divided into sequential 5 minute periods), as well as 5 minutes following each scenario (post-scenario, to observe stress recovery rates). For each participant, the investigators will analyse the participant's root mean square of successive R-R interval differences (rMSSD).
Heart rate variability - pNN50 | During the simulation sessions, throughout the study: 5 minutes at start of each session (Baseline), 5 minutes prior to start of each scenario, for the duration of each scenario (divided into sequential 5 min periods), 5 minutes following each scenario
  As manipulation check, the investigators will compare the team physiological stress scores between the low stress & high stress scenarios by heart rate variability (HRV) monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants HRV will be recorded for 5 minutes at the start of the session (Baseline), 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of each scenario (divided into sequential 5 minute periods), as well as 5 minutes following each scenario (post-scenario, to observe stress recovery rates). For each participant, the investigators will analyse the participant's percentage of successive R-R intervals that differ by more than 50Ms (pNN50).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No